CLINICAL TRIAL: NCT02858206
Title: Prospective, Non-randomised Phase Ⅱ Study of Simultaneous Integrated Boost Radiotherapy and Concurrent Nimotuzumab or Chemotherapy for Locally Advanced Esophageal Carcinoma
Brief Title: Simultaneous Integrated Boost Radiotherapy and Concurrent Nimotuzumab or Chemotherapy for Esophageal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Affiliated Hospital of Hebei University (Other); Beijing Army General Hospital (Other Government); Beijing Hospital (Other Government); Peking University First Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Henan Cancer Hospital (Other Government); The Affiliated Hospital of Inner Mongolia Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zefen Xiao, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-082/1161
Record Dates: First submitted 2016-07-30; First posted 2016-08-08 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Esophageal Neoplasms
Keywords: Locally advanced esophageal cancer; Radiotherapy and nimotuzumab; Concurrent chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — nimotuzumab; Paclitaxel; nedaplatin; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Neoadjuvant nimotuzumab (Experimental): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 4.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively.
  Concurrent nimotuzumab: Patients may receive nimotuzumab 400mg per week which start from 1 week before radiotherapy and in the following 4 weeks after enrollment in the absence of disease progression or unacceptable toxicity.
  Assessment of surgery: Patients eligible for surgery after multiple disciplinary consultation will receive esophagectomy after a 4-6 weeks break after chemoradiation in the absence of any contraindication.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Nimotuzumab; Procedure: Esophagectomy
- Neoadjuvant chemotherapy (Active Comparator): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 4.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively.
  Concurrent chemotherapy: Patients may receive a dosage range of Paclitaxel from 45 to 60 mg/m2 and Nedaplatin 25mg/m2 per week which start from 1 week before radiotherapy and in the following 4 weeks after enrollment in the absence of disease progression or unacceptable toxicity.
  Assessment of surgery: Patients eligible for surgery after multiple disciplinary consultation will receive esophagectomy after a 4-6 weeks break after chemoradiation in the absence of any contraindication.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Paclitaxel; Drug: Nedaplatin; Procedure: Esophagectomy
- Radical nimotuzumab (Experimental): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively.
  Concurrent nimotuzumab: Patients may receive nimotuzumab 400mg per week which start from 1 week before radiotherapy and in the following 4 weeks after enrollment in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Nimotuzumab
- Radical chemotherapy (Active Comparator): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively.
  Concurrent chemotherapy: Patients may receive a dosage range of Paclitaxel from 45 to 60 mg/m2 and Nedaplatin 25mg/m2 per week which start from 1 week before radiotherapy and in the following 4 weeks after enrollment in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Paclitaxel; Drug: Nedaplatin

INTERVENTIONS:
Radiation: IMRT simultaneous integrated boost — To achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively
Drug: Nimotuzumab — nimotuzumab 400mg per week which start from 1 week before radiotherapy and in the following 4 weeks
  Arms: Neoadjuvant nimotuzumab; Radical nimotuzumab
Drug: Paclitaxel — Paclitaxel from 45 to 60 mg/m2 per week which start from 1 week before radiotherapy and in the following 4 weeks
  Other Names: Taxol
  Arms: Neoadjuvant chemotherapy; Radical chemotherapy
Drug: Nedaplatin — Nedaplatin 25mg/m2 per week which start from 1 week before radiotherapy and in the following 4 weeks
  Arms: Neoadjuvant chemotherapy; Radical chemotherapy
Procedure: Esophagectomy — Radical esophagectomy 4-6 weeks after neoadjuvant therapy
  Arms: Neoadjuvant chemotherapy; Neoadjuvant nimotuzumab

SUMMARY:
This prospective, non-randomized phase II study aims to compare radiotherapy and concurrent nimotuzumab with concurrent chemoradiotherapy to obtain a non-inferior pCR rate and pathological lymph node metastases rate in premise of lower toxicities in locally advanced esophageal cancer.

DETAILED DESCRIPTION:
In the era of IMRT and concurrent chemoradiotherapy, the 5-year overall survival of esophageal cancer increase from 10% to about 20%-40%, recurrence rate decrease from 80% to 50%-60%, and local recurrence remains to be the most important type of failure. What called for is to enhance local control without increasing toxicity to improve survival. The investigators have found effective and safe regimen of simultaneously integrated boost radiotherapy in previous study, which can achieve high dose in tumor area with avoid of normal tissues. However, a recent prospective study reported that neoadjuvant chemoradiotherapy resulted in much higher toxicities compares to neoadjuvant chemotherapy (46% vs. 15%, p= 0.04). Although chemoradiotherapy reached a higher pCR rate (28% vs. 9%, p=0.002), patients did not differ in survival in two groups.

Nimotuzumab is an humanized monoclonal antibody against EGFR. Radiotherapy combines Nimotuzumab reveals synergistic effect in head and neck cancers with lower toxicities as compared to concurrent chemoradiotherapy. Our previous study showed that EGFR expression rate were similar in esophageal cancer and head and neck cancers. Based on above results, the investigators design this study which aims to obtain a non-inferior pCR rate and pathological lymph node metastases rate in premise of lower toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinical stage T1-4aN0-1M1a untreated squamous esophageal carcinoma
* KPS≥70
* Adequate organ function
* No known history of drug allergy

Exclusion Criteria:

* Known drug allergy
* Insufficient hepatorenal function
* Severe cardiovascular diseases, diabetes with uncontrolled blood sugar, mental disorders, uncontrolled severe infection, active ulceration which need intervention.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | Up to 1 year
Pathological lymph node metastases rate | Up to 1 year
R0 resection rate | Up to 1 year
Adverse events | Up to 2 years

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Up to 2 years
Overall survival (OS) | Up to 2 years
Recurrence rate | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zefen Xiao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ajani JA, D'Amico TA, Almhanna K, Bentrem DJ, Besh S, Chao J, Das P, Denlinger C, Fanta P, Fuchs CS, Gerdes H, Glasgow RE, Hayman JA, Hochwald S, Hofstetter WL, Ilson DH, Jaroszewski D, Jasperson K, Keswani RN, Kleinberg LR, Korn WM, Leong S, Lockhart AC, Mulcahy MF, Orringer MB, Posey JA, Poultsides GA, Sasson AR, Scott WJ, Strong VE, Varghese TK Jr, Washington MK, Willett CG, Wright CD, Zelman D, McMillian N, Sundar H; National comprehensive cancer network. Esophageal and esophagogastric junction cancers, version 1.2015. J Natl Compr Canc Netw. 2015 Feb;13(2):194-227. doi: 10.6004/jnccn.2015.0028. PMID 25691612
- [Result] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Result] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Result] Kranzfelder M, Schuster T, Geinitz H, Friess H, Buchler P. Meta-analysis of neoadjuvant treatment modalities and definitive non-surgical therapy for oesophageal squamous cell cancer. Br J Surg. 2011 Jun;98(6):768-83. doi: 10.1002/bjs.7455. Epub 2011 Apr 4. PMID 21462364
- [Result] Harari PM, Huang SM. Combining EGFR inhibitors with radiation or chemotherapy: will preclinical studies predict clinical results? Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):976-83. doi: 10.1016/j.ijrobp.2003.09.097. PMID 14967459
- [Result] Ramos-Suzarte M, Lorenzo-Luaces P, Lazo NG, Perez ML, Soriano JL, Gonzalez CE, Hernadez IM, Albuerne YA, Moreno BP, Alvarez ES, Callejo IP, Alert J, Martell JA, Gonzalez YS, Gonzalez YS, Astudillo de la Vega H, Ruiz-Garcia EB, Ramos TC. Treatment of malignant, non-resectable, epithelial origin esophageal tumours with the humanized anti-epidermal growth factor antibody nimotuzumab combined with radiation therapy and chemotherapy. Cancer Biol Ther. 2012 Jun;13(8):600-5. doi: 10.4161/cbt.19849. Epub 2012 Jun 1. PMID 22555809